CLINICAL TRIAL: NCT03723876
Title: Basic Body Awareness Therapy for Persons With Autism. A Pragmatic Randomized Controlled Study
Brief Title: Basic Body Awareness Therapy for Persons With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ingrid Bertilsson
Record Dates: First submitted 2018-06-21; First posted 2018-10-30 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Autism
Keywords: Autism; Movement; Body-mind therapy; Physiotherapy
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Twelve occasions of Basic body awareness therapy, administered once a week, alongside treatment as usual (such as structured everyday support, medicine, contact with social worker).
  Interventions: Behavioral: Body awareness therapy
- Control group (No Intervention): No extra intervention except treatment as usual.

INTERVENTIONS:
Behavioral: Body awareness therapy — The physiotherapist uses body awareness techniques, i.e. guiding the participant in movement qualities such as stability, breathing, flow and grounding. Conscious awareness focused on bodily experiences is a key component to be able to reflect on what your body signals.
  As a baseline a standardized observation of the movement quality of the individual is performed. The physiotherapist needs special education in the body awareness technique used, to rightly perform and analyse the observation and administer the intervention.
  The aim of the body awareness therapy is to raise physical and mental awareness by strengthening the interplay between sensory impressions and motor ability and to gain knowledge of own movement patterns that are not functional and to form alternatives to these.
  Other Names: Basic body awareness therapy
  Arms: Intervention group

SUMMARY:
Autism is a diagnosis with certain criteria, especially social and communicative disabilities. Several body functions may be affected to create these disabilities, such as lack of ability to understand that other people think or feel differently than the person with autism, difficulty to experience bodily signals or deviant function of sensory modalities.

Several theories describe that our physical, physiological, psychological and existential being can not be separated from each other. The combination of described difficulties in autism makes the perception of the surrounding world or the people within it difficult to understand or interpret, i.e., lack of a sense of coherence. The inner experience of the person as well as the expression of his/her movement qualities will be the effects.

There are physiotherapeutic intervention techniques of body awareness, with the purpose to increase the connection to the body and to work with more functional movements. Instead of working with improving the well-being by cognitive top-down techniques, body awareness techniques work bottom-up.

The hypothesis is that an intervention with body awareness therapy will increase the possibility for persons with autism to improve movement quality, and increase contact with bodily signals. It will give a better chance to understand and interpret the world and people in different context, conquering a sense of coherence.

The study include at least 40 participants with autism randomized to two groups: 1.) intervention once a week for 12 weeks and 2. ) a control group (who will be invited to the therapy after ending study participation). They will be recruited from patient records in habilitation care. The criteria are: having autism, being 15-30 years, not having an intellectual impairment and not having a severe depression. The participants are to have been assessed with the standardized "Basic Body Awareness Scale Movement Quality and Experience", BAS MQ-E, and been found to being relevant participants for body awareness intervention in regard to the expressed individual health problem.

Two assessments will be used. The primary one addresses each participants´s individual health problem, using a visual 11-graded scale (NRS), grading the present experience of the health problem. The secondary one is BAS MQ-E. The assessments will be administered as follows: i) prior to; NRS + BAS MQ-E, ii) after 7 occasions; NRS and iii) maximum 2 months after intervention; NRS + BAS MQ-E.

DETAILED DESCRIPTION:
Introduction Movement quality is a concept that describes how movements are performed in space, time and amount of energy. When the quality is good, the movement is perceived as unrestricted and gives a sense of freedom, physically and mentally. Movement quality and body awareness are dependent on each other. Body awareness is the ability to be consciously present and interpret signals from your own body. A physiotherapeutic treatment method that describes how movement quality and body awareness interact on a deeper level is Basic Body Awareness Therapy (BBAT).

The purpose of BBAT is to raise physical and mental awareness by strengthening the interplay between sensory impressions and motor ability, gaining knowledge of movement patterns and habits that are not functional. Man's ability to perceive, take care of, control and use the body in a functional manner affects the quality and expression of the movements. According to the theory behind BBAT, movement quality and body awareness are both important abilities to develop bodily self-consciousness.

In order to distinguish between oneself and others, ability to gather and make conscious sensory impressions through the body is demanded. In order to understand the impressions and the world around us, one need to be able to integrate sensory impressions to each other into an information with deeper meaning, the creation of perceptual coherence. The perceptual coherence is the basis for knowledge of one's own body and movement quality. Body awareness increases with more experience of movement. based on the physiotherapeutic bodyself, the subjective ("I as my body") and objective ("I in my body") identity we use to meet and understand the world. The bodyself comes to expression through the degree of movement quality and can as such be observed.

When people with autism grow up, their development differs from typically developed peers. They may find it difficult to understand that other people have their own thoughts and feelings, so-called theory of mind and to understand their own feelings and inner states. They may lack central coherence, being able to merge details to the whole. They may also react differently to smells, flavors, sounds or materials carried on the body, having difficulty imitating others, have less flexibility to achieve motion targets, have poorer motor skills and/or sensorimotor function. In autism, the ability for multi-sensory integration is often inadequate. In this way, context and meaning can become less comprehensible and meaningful. This can lead to changes in the bodyself.

As children with autism exhibit worse body awareness and movement quality than children with typical development, it may be likely that body and movement experiences are reduced through upbringing. This can affect physical and mental health, as seen in autism. A study from 1991 examined how young adults with autism describe how movement quality from a body function perspective affects their ability to maintain daily activities and participation. The attention it required of the individual to attempt to master stereotyped movements to be considered "normal", resulted in increased mental energy utilization as they constantly watched their own behavior, also creating anxiety. In a previous study we interviewed eleven young adults with autism about their experiences about body and movement, as well as examined them with one motor and one body awareness instrument. The results showed conflicting feelings about their bodies and movements, but also how movement quality was related to the way the individual had access to functional strategies to handle everyday situations or not. There is little knowledge about the effects of various interventions that focus on body awareness and movement quality in this group.

The objective of this study is to investigate effects of a BBAT intervention for young adults with autism. Research question: Can an intervention with BBAT help young adults with autism to improve their movement qualities in everyday activities and achieve individually expressed need to improve?

Participants The participants will be young adults with autism, living in the region of Skaraborg in Västra Götaland or in the region of Kronoberg. See 10. Eligibility criteria.

All patients with autism, within the criteria, that has been examined with BAS MQ-E may be eligible for participation in this study. Individual needs for improvement are discussed with each individual. If relevant needs are expressed, which may be encountered with BBAT, and the patient is motivated for intervention, he/she will be included in the study following informed consent. The expressed individual need will be defined in a statement, such as "I experience muscle tensions" or "I can calm myself before bedtime". The intervention will start within one month after performing BAS MQ-E and administered individually. A control group is used within the patient group. With a significance level of 0.05, a power of 0.8 and a moderate effect, at least 20 participants are calculated for in the intervention and control groups respectively.

Ethics The study is approved by The Regional ethical review board in Gothenburg (Dnr 651-17).

Instruments Numeric rating scale Individually expressed health problem is estimated on an individualized 11-degree numeric rating scale (NRS). See 9. Outcome measures.

BAS MQ-E Movement quality will be examined with Body Awareness Scale Movement Quality and Experience (BAS MQ-E). See 9. Outcome measures.

Methods A pragmatic randomized controlled study, pRCT, will be conducted. Participants are jointly managed for Skaraborg and Kronoberg and randomized to intervention group and control group. The distribution is managed by an independent person. Randomization takes place by using a random generator function at http://gallerit.se/slumptal/, with numbers 1 and 2. All 1 means that the participant is randomized to the intervention group, all 2 to the control group.

Intervention group: The layout is individualized based on the results of BAS MQ-E, all three parts. The individually expressed health problem is estimated on the NRS scale. After assessment, 12 occasions are given with BBAT approximately once a week (3-4 months).

Control group: Treatment as usual for 3-4 months. Individualized NRS estimation and assessment with BAS MQ-E are performed according to flowchart. The participant will then have access to BBAT if they wish.

Data collection BAS MQ-E (1) used in the study has been collected either from a previous validation study or from everyday clinic. BAS MQ-E (2), parts Movement test and Questionnaire, will be performed maximum 1 month after the end of the intervention by an independent examiner. Own rating of the individualized health problem using the VAS will be performed prior to the intervention (1), after 7 occasions of intervention (2) and maximum 2 months after last occasion of intervention at 12 weeks, approximately 20 weeks total (3).

Data analysis The primary outcome measure are the results from the NRS ratings. Further, the scores from BAS MQ-E, parts Movement test and Questionnaire, as secondary outcome measure. ANOVA will be used for statistical analysis of differences for repeated measures prior to, during and after the intervention. The intervention- and control groups will be analyzed to each other for any statistical significant difference using Mann Whitney U test (significance level p<0,05).

Clinical significance of the study Body and movements are often described as problems in persons with autism. But it omits that there are also resources in the body to find strategies for everyday life. By strengthening body functions and enhancing movement quality and body awareness through a body therapy intervention, the person with autism can better understand themselves. Strengthened body functions then provide the basis for the individual's opportunities for development and increased participation in society. Expected results thus follow the UN Convention on the Rights of Persons with Disabilities, i.e. to eliminate obstacles for people with disabilities to enjoy their human rights and participation, in full and equal to others.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with an autism diagnosis (F84* in ICD-10)
* 15-30 years
* accepted for care at habilitation unit

Exclusion Criteria:

* diagnosed with intellectual disability (F70*-F73*, F78*-F79* in ICD-10)
* medium or severe depression
* major problems with country´s native language

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change of experienced health problem from Numeric rating scale | 1.) Maximum 2 months prior to intervention, 2.) after 7 occasions of therapy and 3.) maximum 2 months after last occasion of intervention at 12 weeks, approximately 20 weeks total
  The scale is a Numeric rating scale, 15 cm long with 11 vertical lines, marked from 0 to 10. One individual health problem will be identified by the participant. The health problem needs to be judged by the physiotherapist as relevant to meet with body awareness intervention. If so, the sentence will be typed above the scale before rating. A health problem could for instance be "I experience muscle tensions". 0=no problems experienced and 10=extreme problems, i.e. 0 is the best value. In order to follow any process of change, an intermediate measure will be performed.

SECONDARY OUTCOMES:
Change of results of Body Awareness Scale Movement Quality and Experiences, BAS MQ-E | 1.) Maximum 2 months prior to intervention and 2.) maximum 2 months after last occasion of intervention at 12 weeks, approximately 20 weeks total
  1.) Movement test: 23-item physiotherapeutic observation of movement quality, rated ordinally in a 5-graded scale, 0=vitality to 4=pathology/not executing. 2.) Questionnaire: Own rating of 7 items about how one´s body works in everyday life, 4-graded ordinally scale, 0=no problems to 3=don´t work 3.) Experienced-based interview: The participant is asked to describe experiences from his/her body during four standardized movements from the Movement test (part one). Their descriptions are written down verbatim. Both qualitative and quantitative data are obtained with this instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Sjödahl Hammarlund, As.professo, Study Chair — Lund University
Locations (2):
- Sweden (2):
  - Vuxenhabiliteringen, Vaxjo, Kronoberg County
  - Habiliteringen Vastra Gotalandsregionen, Skövde, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertilsson I, Gyllensten AL, Opheim A, Gard G, Sjodahl Hammarlund C. Understanding one's body and movements from the perspective of young adults with autism: A mixed-methods study. Res Dev Disabil. 2018 Jul;78:44-54. doi: 10.1016/j.ridd.2018.05.002. Epub 2018 May 15. PMID 29772450
- [Background] Bhat AN, Landa RJ, Galloway JC. Current perspectives on motor functioning in infants, children, and adults with autism spectrum disorders. Phys Ther. 2011 Jul;91(7):1116-29. doi: 10.2522/ptj.20100294. Epub 2011 May 5. PMID 21546566
- [Background] Cesaroni L, Garber M. Exploring the experience of autism through firsthand accounts. J Autism Dev Disord. 1991 Sep;21(3):303-13. doi: 10.1007/BF02207327. PMID 1938776
- [Background] Einspieler C, Sigafoos J, Bolte S, Bratl-Pokorny KD, Landa R, Marschik PB. Highlighting the first 5 months of life: General movements in infants later diagnosed with autism spectrum disorder or Rett Syndrome. Res Autism Spectr Disord. 2014 Mar;8(3):286-291. doi: 10.1016/j.rasd.2013.12.013. Epub 2014 Jan 9. PMID 29770159
- [Background] Frith U, Happe F. Autism: beyond "theory of mind". Cognition. 1994 Apr-Jun;50(1-3):115-32. doi: 10.1016/0010-0277(94)90024-8. PMID 8039356
- [Background] Gyllensten, A. L. (2012). Basal kroppskännedom. i G. Biguet, R. Keskinen-Rosenqvist, & A. Levy Berg, Att förstå kroppens signaler - sjukgymnastiska perspektiv (ss. 189-206). Lund: Studentlitteratur.
- [Background] Gyllensten, A. L., Hansson, L., & Ekdahl, C. (2003). Patient experiences of basic body awareness therapy and the relationship with the physiotherapist. Journal of Bodywork and Movement Therapies, 7, 173-183.
- [Background] Hedlund, L. (2014). Basal kroppskännedom och psykomotorisk funktion hos personer med allvarlig psykisk sjukdom. Doctoral thesis, Lund: Department of Health Science, Division of Physiotherapy.
- [Background] Kopp S, Beckung E, Gillberg C. Developmental coordination disorder and other motor control problems in girls with autism spectrum disorder and/or attention-deficit/hyperactivity disorder. Res Dev Disabil. 2010 Mar-Apr;31(2):350-61. doi: 10.1016/j.ridd.2009.09.017. Epub 2009 Nov 11. PMID 19910158
- [Background] Lai MC, Lombardo MV, Baron-Cohen S. Autism. Lancet. 2014 Mar 8;383(9920):896-910. doi: 10.1016/S0140-6736(13)61539-1. Epub 2013 Sep 26. PMID 24074734
- [Background] Norman, G., & Streiner, D. (2014). Biostatistics. The bare essentials. Ontario: PMPH-USA Limited.
- [Background] Regeringskansliet. (2008). FN:s konvention om rättigheter för personer med funktionsnedsättning. Hämtat från http://www.regeringen.se/contentassets/0b52fa83450445aebbf88827ec3eecb8/fns-konvention-om-rattigheter-for-personer-med-funktionsnedsattning-ds-200823
- [Background] Rizzolatti G, Fabbri-Destro M. Mirror neurons: from discovery to autism. Exp Brain Res. 2010 Jan;200(3-4):223-37. doi: 10.1007/s00221-009-2002-3. Epub 2009 Sep 18. No abstract available. PMID 19760408
- [Background] Simons J, Leitschuh C, Raymaekers A, Vandenbussche I. Body awareness in preschool children with psychiatric disorder. Res Dev Disabil. 2011 Sep-Oct;32(5):1623-30. doi: 10.1016/j.ridd.2011.02.011. Epub 2011 Mar 24. PMID 21435833
- [Background] Skjaerven, L., Gard, G., & Kristoffersen, K. (2003). Basic elements and dimensions to the phenomenon of quality of movement - a case study. Journal of bodywork and movement therapies.
- [Background] Whyatt C, Craig C. Sensory-motor problems in Autism. Front Integr Neurosci. 2013 Jul 18;7:51. doi: 10.3389/fnint.2013.00051. eCollection 2013. PMID 23882194